CLINICAL TRIAL: NCT06094985
Title: Prognostic Markers for a Better Follow-up in Head and Neck Cancer.
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Näsman, Assoc Prof, Karolinska Institutet
Other Study IDs: 2023-04222-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — DNA extracted from tumour and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with head and neck cancer: Patient diagnosed with head and neck cancer
  Interventions: Genetic: DNA exome sequencing of tumor and blood

INTERVENTIONS:
Genetic: DNA exome sequencing of tumor and blood — A piece from tumor and a blood sample will be collected during surgery. DNA will be extracted and presence of tumor specific mutations/aberrations will be analysed with a DNA exome seq panel. Presence of identified markers will be followed in blood samples with the same panel and these blood samples will be collected in routine follow-up during the first two years. Presence of markers over time in blood will be correlated to outcomes 1-5.

SUMMARY:
To identify tumor specific DNA mutations and aberrations and to follow these in blood over time to predict treatment response/survival and secondly to correlate presence of these markers in blood to pathological parameters (LVI, Pn, WPOI and margins), radiological findings and to tumor stage.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with head and neck cancer
* Treatment includes surgery
* Consent to participate

Exclusion Criteria:

* No consent
* Age below 18 years
* No surgery
* No tumor material to sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with a primary head and neck cancer Nov 2023 to May 2024 at Karolinska will be asked to participate.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-02-12 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 2 years
  Recurrent disease within 2 years after surgery. Is presence of these DNA changes in blood correlated to recurrence?
Survival | 2 years
  Alive/dead. Is presence of these DNA changes in blood correlated to survival?
Treatment response | 6 months
  Is presence of these DNA changes in blood correlated to treatment response?

SECONDARY OUTCOMES:
Pathological parameters | 6 months
  Is presence of these DNA changes correlated to pathological parameters (LVI, Pn, WPOI and margins).
Radiological parameters | 9 months
  Is presence of these DNA markers in blood correlated to PET-findings?
Stage | 2 years
  If patients are stratified by stage, are there any differences in Outcome 1-5 (please see above)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Näsman, MD PhD, Principal Investigator — Karolinska institutet and Karolinska Universitetssjukhuset
Locations (1):
- Karolinska universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided